CLINICAL TRIAL: NCT06030154
Title: Developing and Evaluating a Positive Valence Treatment for Alcohol Use Disorder With Anxiety or Depression
Brief Title: Amplification of Positivity for Alcohol Use
Acronym: AMP-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: University of California, San Diego (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-003; R34AA030688 (NIH)
Record Dates: First submitted 2023-07-12; First posted 2023-09-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Anxiety; Depression
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amplification of Positivity Therapy (Experimental): AMP-A will involve 12, one-hour weekly therapy sessions completed one-on-one with a therapist. The sessions and between-session homework will focus on amplifying positive thoughts, emotions, and behaviors to address anxiety/depression and alcohol use.
  Interventions: Behavioral: Amplification of Positivity Therapy; Behavioral: Surveys and Interviews
- Cognitive Behavioral Therapy (Active Comparator): The CBT intervention will involve 12, one-hour weekly therapy sessions completed one-on-one with a therapist. The sessions and between-session homework will focus on monitoring of the relationship between thoughts, emotions, and alcohol use.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Surveys and Interviews

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy
Behavioral: Amplification of Positivity Therapy — Amplification of Positivity Therapy
  Arms: Amplification of Positivity Therapy
Behavioral: Surveys and Interviews — Participants will answer questions regarding their mental and physical health as well as their substance use on the computer and in an interview format.

SUMMARY:
The proposed study consists of two phases. During Phase 1, the investigators will recruit a small sample of participants to complete a psychosocial intervention termed Amplification of Positivity (AMP) for individuals experiencing comorbid depression or anxiety disorders and alcohol use disorder (AMP-A). These participants will be asked to provide both qualitative and quantitative input about the AMP-A intervention. Based on their input and clinician input, the AMP-A manual will be modified for use in Phase 2. The goal is to recruit up to 20 participants in order to ensure there will be at least 8 participants who complete all sessions of AMP-A. Phase 2 is a randomized clinical trial (RCT) protocol in which individuals experiencing comorbid depression or anxiety disorders and alcohol use disorder will be randomized to complete AMP-A or an evidence-based cognitive-behavioral therapy (CBT) intervention. Up to 100 participants will be recruited in order to reach a target of N=60. Assessed outcomes will include participant acceptability and completion rates, participant compliance with the intervention, positive and negative affect, substance use- and depression and anxiety-related symptom severity, functional disability, and neural reactivity to reward and alcohol cues during functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Substance use disorder, including alcohol use disorder, is characterized by enhanced neural responsivity to drug (alcohol) cues, but reduced neural responsivity to non-drug reward cues. These effects may be exacerbated by comorbid major depressive disorder (MDD) or symptoms of anhedonia, comorbidities which are particularly high amongst alcohol use disorder. Response rates for current interventions with alcohol use disorder are rather poor, with only 58% experiencing benefits greater than control conditions. There is a need to identify interventions that may target reward responsivity in a way that would promote recovery, reduce affective disturbance, and support better long-term functioning for individuals experiencing alcohol use disorder and comorbid depression and anxiety disorders. Positive affect interventions have recently been developed and tested in other populations (i.e., HIV, anxiety/depression) as a way of enhancing positive valence and reward processing. These interventions have shown significant promise in these populations but have yet to be examined in the context of alcohol use disorder.

The current study would test the feasibility and acceptability of a 12-session protocol focused on amplification of positivity with populations experiencing comorbid alcohol use disorder and depression or anxiety disorders and explore the impact of the intervention on positive affect, negative affect, alcohol use and craving, and neural response patterns during reward and drug cue processing. The proposed project would support the final stages of intervention development. First, an initial pilot study will be conducted to obtain qualitative and quantitative input from N=8 participants with Alcohol Use Disorder (AUD) + Anxiety/Depression (ANX/DEP) who are asked to engage in the amplification of positivity for AUD intervention (AMP-A) and their clinicians to inform modifications to the AMP-A manual. Then, a pilot randomized clinical trial (RCT) will be conducted in which N=60 individuals with Alcohol Use Disorder (AUD) + Anxiety/Depression (ANX/DEP) will be randomized to complete the modified AMP-A intervention or a cognitive behavioral therapy (CBT)intervention. Intervention will consist of 12 sessions that may be done virtually or in-person. Participation in both phases will include completion of interview-based and self-report measures at pre-treatment, weekly during treatment, at post-treatment, and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Meeting diagnostic criteria for alcohol use disorder 42 according to the DSM-5.
3. Reports that they would like to seek treatment for AUD and that AUD is one of the primary challenges they would like to address in treatment.
4. Phase 1: Significant depression or anxiety symptoms as indexed by scoring Patient Health Questionnaire (PHQ-9) ≥ 10 and/or Overall Anxiety Severity and Impairment Scale (OASIS) ≥ 8. Phase 2: Significant depression or anxiety symptoms as indexed by scoring ≥ 55 on either of the NIH PROMIS ((Patient-Reported Outcomes Measurement Information System) Depression and/or Anxiety scales.
5. Below normative levels of positive affect as indexed by PROMIS Positive Affect <50.
6. Able to provide written informed consent.
7. Have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. Unwillingness or inability to complete any of the major aspects of the study protocol, including self-report or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task). In addition, the neuroimaging portion of the protocol will be optional.
2. Non-correctable vision or hearing problems that interfere with the participant's ability to complete study assessments.
3. No telephone or easy access to telephone.
4. Diagnosis of Schizophrenia spectrum, other psychotic disorders, obsessive-compulsive disorder, eating disorders, substance use disorders within the past year other than alcohol use disorder or cannabis use disorder, or bipolar I disorder. Mild binge eating disorder will be considered for inclusion on a case-by-case basis at the discretion of the PI.
5. Active suicidal ideation with plan and intent to attempt suicide within the next month.
6. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
7. A positive test for drugs of abuse, including alcohol (breath test) and substances of dependence that are not physician prescribed (i.e., cocaine, cannabis, opioids, stimulants).at the time of baseline assessments. Participants will be asked to refrain from using alcohol within 24 hours prior to assessment sessions and to refrain from using marijuana within 48 hours of assessment sessions.
8. Current use of a medication within the 6 weeks prior to enrolling in the study that could potentially affect brain functioning and/or the positive valence system (e.g., anxiolytics, antipsychotics, mood stabilizers, opioid antagonists such as naltrexone or other medications specifically targeting alcohol use or cravings). The current use of antidepressants (i.e., SSRIs), benzodiazepines, and psychostimulants will not be excluded as long as the dose has remained consistent for 6 weeks prior to baseline assessment sessions. Individuals who are on stable doses (≥ 6 weeks) of mood stabilizers or antipsychotics may be included if it is determined that they are being prescribed for purposes of treating unipolar depression or anxiety. Inclusion of individuals reporting other types of medications or supplements not listed or considered this far will be at the discretion of the PI according to evidence in the literature of it affecting brain function or brain blood flow.
9. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, and excessive caffeine intake > 1000 mg/day) - Phase 2 only
10. Concurrent engagement in psychosocial treatments that specifically target alcohol use disorder or mood/anxiety symptoms and began within 12 weeks of baseline assessments. Individuals concurrently receiving psychosocial treatments for other symptoms, or that are not specifically targeting symptoms (e.g., ongoing support groups) will not be excluded as long as the dose of treatment (i.e., frequency of sessions) has not changed significantly within 6 weeks prior to enrolling in the study.
11. MRI contraindications (for those in Phase 2 opting into this portion) including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy - Phase 2 only
12. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider).
13. Severity of alcohol use disorder requiring more intensive treatment (i.e., intensive outpatient or residential), as determined by licensed clinician determination of American Society of Addiction Medicine (ASAM) Criteria ≥ 0-1 across dimensions, with the exception of a '2' on the emotional dimension.
14. Given the current study involves development of the positive affect intervention, we will not enroll any special vulnerable populations (pregnant women, fetuses, neonates, prisoners, children).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Perceived acceptability and satisfaction of the intervention as measured with the Adherence and Acceptability Scale (AAS) | Average of total scores from the following time points: pre-treatment, 2 weeks after starting treatment, 6 weeks after starting treatment, and at post-treatment (average of 16 weeks after baseline assessment)
  This measure assesses the acceptability and tolerability of the intervention and is the primary outcome for Phase 1. Scores may range from 10 to 70, with higher scores indicating greater acceptability of treatment and greater anticipated ability to adhere to it.
Change in positive affect self-report measured with National Institute of Health (NIH) Patient Reported Outcome Measurement and Information System (PROMIS) Positive Affect score | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  National Institute of Health (NIH) Patient Reported Outcome Measurement and Information System (PROMIS) Positive Affect Scale, which is reported as a T score. The score is presented as a T score with a mean of 50 and a standard deviation of 10, with a range of 0-100. Higher scores indicate greater positive affect or better outcome. This is a primary outcome for Phase 2.
Change in number of drinking days in the past month | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  As measured through self-reported drinking days using Timeline Followback. This is a primary outcome for Phase 2.

SECONDARY OUTCOMES:
Distress/Endorsement Validation Scale (DEVS) | Average of total scores from the following time points:2 weeks after starting treatment, post-treatment (average of 16 weeks after baseline assessment)
  This measure assesses two factors, distress (7 items) and endorsement (3 items) and is a secondary outcome for Phase 1. The distress subscale score ranges from 7 to 63, with higher scores indicating more distress experienced during the intervention. The endorsement subscale ranges from 3 to 27, with higher scores indicating greater endorsement of the intervention.
Change in Average drinks per drinking day | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  As measured through self-reported drinks using a Timeline Followback interview. This is a secondary outcome for Phase 2.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  This measure assesses symptoms of anxiety over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with a range of 0-100. Higher scores indicating greater symptoms of anxiety. This is a secondary outcome for Phase 2.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  This measure assesses symptoms of depression over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with a range of 0-100. Higher scores indicating greater symptoms of depression. This is a secondary outcome for Phase 2.
Change in Sheehan Disability Scale (SDS) | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  This measure assesses functional impairment, with higher scores indicating greater disability. Scores range from 0 to 30. This is a secondary outcome for Phase 2.
Change in the NIH Toolbox Loneliness survey | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  This measure assesses feelings related to loneliness over the past month. The total score ranges from 5-25, with higher scores indicating greater feelings of loneliness. This is a secondary outcome for Phase 2.
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Meaning and Purpose Scale | Trajectory of change from pre-treatment to post-treatment (last time point assessed on average 16 weeks after baseline assessment)
  This measure assesses general feelings related to meaning and purpose in one's life. The score is presented as a T score with a mean of 50 and standard deviation of 10 with a range of 0-100. Higher scores indicating greater feelings of meaning and purpose. This is a secondary outcome for Phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Aupperle, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan on sharing human data from the completed project with qualified investigators via the National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAADA) in compliance with NOT-AA-22-011 as applicable.
Supporting Information: Study Protocol
Time Frame: Within 6 months of the start of the award, the investigators will complete the Data Submission Agreement and Data Expected aspects of this project within NIAAADA, with the first project data uploaded to NDA within one year of the start of the award, in accordance with applicable Data Sharing Terms and Conditions of the award. The investigators will perform QA/QC checks on data within 4 months after the submission due date and address any identified issues. Data will then be cumulatively every 6 months throughout the project.

REFERENCES:
- [Background] Akeman E, White E, Wolitzky-Taylor K, Santiago J, McDermott TJ, DeVille DC, Stewart JL, Paulus M, Taylor CT, Aupperle RL. Amplification of Positivity Therapy for Co-occurring Alcohol Use Disorder with Depression and Anxiety Symptoms: Pilot Feasibility Study and Case Series. Behav Modif. 2022 Sep;46(5):1021-1046. doi: 10.1177/01454455211030506. Epub 2021 Jul 12. PMID 34253077
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463
- [Background] Kryza-Lacombe M, Pearson N, Lyubomirsky S, Stein MB, Wiggins JL, Taylor CT. Changes in neural reward processing following Amplification of Positivity treatment for depression and anxiety: Preliminary findings from a randomized waitlist controlled trial. Behav Res Ther. 2021 Jul;142:103860. doi: 10.1016/j.brat.2021.103860. Epub 2021 Apr 15. PMID 33894554

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT06030154/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT06030154/ICF_001.pdf